CLINICAL TRIAL: NCT06211764
Title: A Phase 3, Randomized, Open-label, Multi-center Study Evaluating the Efficacy and Safety of TAR-200 Versus Investigator's Choice of Intravesical Chemotherapy in Participants Who Received Bacillus Calmette-Guérin (BCG) and Recurred With High-risk Non-muscle-invasive Bladder Cancer (HR-NMIBC) and Who Are Ineligible for or Elected Not to Undergo Radical Cystectomy
Brief Title: A Study of TAR-200 Versus Intravesical Chemotherapy in Participants With Recurrent High-Risk Non-Muscle-Invasive Bladder Cancer (HR-NMIBC) After Bacillus Calmette-Guérin (BCG)
Acronym: SunRISe-5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17000139BLC3004; 17000139BLC3004 (Other: Janssen Research & Development, LLC); 2023-507685-10-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Neoplasms
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: TAR-200 (Experimental): Participants will receive intravesical TAR-200 every 3 weeks during an induction phase and every 12 weeks during a maintenance phase.
  Interventions: Drug: TAR-200
- Group B: Mitomycin C (MMC) or Gemcitabine (Active Comparator): Participants will receive either single agent intravesical MMC or gemcitabine every week during an induction phase and every 4 weeks during a maintenance phase.
  Interventions: Drug: Mitomycin C; Drug: Gemcitabine

INTERVENTIONS:
Drug: TAR-200 — Participants will receive TAR-200 intravesically.
  Other Names: JNJ-17000139
  Arms: Group A: TAR-200
Drug: Mitomycin C — Participants will receive MMC intravesically.
  Arms: Group B: Mitomycin C (MMC) or Gemcitabine
Drug: Gemcitabine — Participants will receive gemcitabine intravesically.
  Arms: Group B: Mitomycin C (MMC) or Gemcitabine

SUMMARY:
The purpose of this study is to compare disease free survival (DFS) in participants with recurrence of papillary-only high-risk non-muscle-invasive bladder cancer (HR-NMIBC) within 1 year of last dose of Bacillus Calmette-Guérin (BCG) therapy and who refused or are unfit for Radical Cystectomy (RC), receiving TAR-200 versus investigator's choice of single agent intravesical chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis by local pathology (within 90 days of documented informed consent) of recurrent, papillary-only high-risk non-muscle-invasive bladder cancer (HR-NMIBC) [defined as high-grade Ta or any T1, no carcinoma in situ (CIS)]
* Participants with variant histologic subtypes are allowed if tumor(s) demonstrate urothelial (transitional cell histology) predominance. However, neuroendocrine, and small cell variants will be excluded
* Participants must be ineligible for or have elected not to undergo Radical Cystectomy (RC)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status Grade of 0, 1, or 2

Exclusion Criteria:

* Presence of CIS at any point from time of diagnosis of papillary-only HR-NMIBC recurrence to randomization. Additionally, presence or history of histologically confirmed, muscle-invasive, locally advanced, nonresectable, or metastatic urothelial carcinoma (that is, T2, T3, T4, N+, and/or M+)
* Presence of any bladder or urethral anatomic feature that, in the opinion of the Investigator, may prevent the safe placement, indwelling use, or removal of TAR-200. Participants with tumors involving the prostatic urethra in men will be excluded
* A history of clinically significant polyuria with recorded 24-hour urine volumes greater than 4000 milliliters (>4000 mL)
* Indwelling catheters are not permitted; however, intermittent catheterization is acceptable
* Previous treatment with TAR-200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2030-11-27 (Estimated); Study Completion 2031-04-14 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 6 years 7 months
  DFS will be measured as the time from randomization to the time of the first recurrence of high-risk non-muscle-invasive bladder cancer (HR-NMIBC) [high grade (HG) Ta, any T1 or carcinoma in situ (CIS)], progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 6 years 7 months
  RFS will be measured as the time from randomization to the time of the first recurrence of HR-NMIBC (HG Ta, any T1 or CIS), or death due to any cause, whichever occurs first.
Time to Next Intervention (TTNI) | Up to 6 years 7 months
  TTNI will be measured as the time from randomization to the time of next intervention (localized or systemic) for the treatment of bladder cancer.
Time to Disease Worsening (TTDW) | Up to 6 years 7 months
  TTDW is measured as the time from randomization to cystectomy, systemic therapy, or radiation therapy (treatments of disease worsening).
Time to Progression (TTP) | Up to 6 years 7 months
  TTP will be measured as the time from randomization to the time of first documented evidence of disease progression (that is, progression to muscle-invasive bladder cancer [MIBC] [T greater than or equal to {>=} 2], lymph node disease [N+], or distant disease [M+]), or death due to disease progression, whichever occurs first.
Overall Survival (OS) | Up to 6 years 7 months
  OS is defined as the time from randomization to death, due to any cause.
DFS Rate at 12 and 24 Months | At 12 and 24 months
  DFS rate that is percentage of participants with DFS at 12 and 24 months will be reported.
Number of Participants with Adverse Events (AEs) According to Common Terminology Criteria for Adverse Events (CTCAE) | Up to 6 years 7 months
  Number of participants with AEs by severity grade as assessed by CTCAE version 5 will be reported. Grade refers to the severity of AE as follows: Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening; Grade 5- Death related to adverse event.
Number of Participants With Change from Baseline in Laboratory Abnormalities | Up to 6 years 7 months
  Number of participants with change from baseline in laboratory abnormalities (including hematology, clinical chemistry and routine urinalysis) will be reported.
Number of Participants With Change from Baseline in Vital Signs Abnormalities | Up to 6 years 7 months
  Number of participants with change from baseline in vital signs including temperature, pulse/heart rate, respiratory rate, and blood pressure (systolic and diastolic) (supine) will be reported.
Change from Baseline in European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire (EORTC QLQ) - C30 Scores | Up to 5 years
  EORTC QLQ-C30 is a 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. It includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea or vomiting), and a global health status or HRQoL scale. Ratings for each item range from 1 (not at all) to 4 (very much).
Change from Baseline in EORTC QLQ- Non-Muscle-Invasive Bladder Cancer (NMIBC) 24 Scores | Up to 5 years
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with NMIBC. The questionnaire is designed to supplement the QLQ-C30 and incorporates 6 multi-item scales (urinary symptoms, malaise, future worries, bloating and flatulence, sexual function and male sexual problems) and 5 single items (intravesical treatment issues, sexual intimacy, worries about risk of contaminating partner, sexual enjoyment, and female sexual problems). Ratings for each item range from 1 (not at all) to 4 (very much).
Proportion of Participants With Meaningful Change in EORTC QLQ-C30 and EORTC QLQ-NMIBC24 Scores | Up to 5 years
  Proportion of participants with meaningful change in EORTC QLQ-C30 and EORTC QLQ-NMIBC24 scores will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (123):
- United States (29):
  - Arkansas Urology, Little Rock, Arkansas
  - Genesis Research LLC, Los Alamitos, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - University of California San Francisco, San Francisco, California
  - Genesis Research LLC, Torrance, California
  - Colorado Clinical Research, Lakewood, Colorado
  - Florida Urology Partners, Riverview, Florida
  - Northwestern University, Chicago, Illinois
  - UroPartners, Chicago Ridge, Illinois
  - Urology of Indiana, Carmel, Indiana
  - First Urology, PSC, Jeffersonville, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - Comprehensive Urology, Royal Oak, Michigan
  - Specialty Clinical Research of St Louis, St Louis, Missouri
  - Associated Medical Professionals, Syracuse, New York
  - The Urology Group, Cincinnati, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Centers for Advanced Urology LLC d b a MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Low Country Urology Clinics, North Charleston, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Spokane Urology, Spokane, Washington
- Argentina (5):
  - Clinica Santa Isabel, Buenos Aires
  - Investigaciones Clinico Moleculares (ICM), CABA
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Hospital Privado de la Comunidad, Mar del Plata
- Belgium (5):
  - AZ Sint-Jan, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - Algemeen ziekenhuis Maria Middelares, Ghent
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (9):
  - Fundacao Pio XII, Barretos
  - NAIC Nair Antunes Instituto do Cancer, Bauru
  - Hospital das Clinicas da Universidade Estadual de Campinas UNICAMP, Campinas
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital da Bahia, Salvador
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- China (10):
  - Peking University First Hospital, Beijing
  - West China School of Medicine/West China Hospital, Sichuan University, Cheng Du Shi
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Shengjing Hospital Of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The Second Hospital Of Tianjin Medical University, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Medical College of Huazhong University Science Technology of Medicine Health Management, Wuhan
  - Xi an Jiaotong University Hospital, Xi'an
- France (7):
  - Hopital Claude Huriez, Lille
  - Polyclinique de Limoges - Francois Chenieux, Limoges
  - Institut Paoli Calmettes, Marseille
  - APHP - Hopital Bichat - Claude Bernard, Paris
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Hopital Foch, Suresnes
- Germany (6):
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Halle Saale, Halle
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Urologie Neandertal Praxis Mettmann, Mettmann
  - Klinikum der Universitaet Muenchen, München
- Italy (9):
  - Ospedale San Donato, Arezzo
  - Ospedale Provinciale di Macerata, Macerata
  - San Raffaele Hospital, Milan
  - Istituto Dei Tumori Di Milano, Milan
  - Ospedale S. Maria Delle Croci, Ravenna
  - Universita Campus Bio-Medico di Roma, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Clinico Humanitas, Rozzano
  - PO Molinette Azienda Ospedaliero Universitaria Citta della Salute e della Scienza di Torino, Torino
- Japan (8):
  - Funabashi Municipal Medical Center, Funabashi Shi
  - Hakodate Goryoukaku Hospital, Hakodate
  - Hyogo Prefectural Amagasaki General Medical Center, Hyōgo
  - Niigata Cancer Center Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Toho University Sakura Medical Center, Sakura
  - Toranomon Hospital, Tokyo
  - Yokohama City University Medical Center, Yokohama
- Poland (9):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - IN VIVO Sp. z o.o, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersytecki Szpital Kliniczny nr 4, Lublin
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Szpital Wojewodzki im Sw Lukasza SP ZOZ, Tarnów
  - MICS Centrum Medyczne Torun, Torun
  - Mazowiecki Szpital Onkologiczny, Wieliszew
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Romania (5):
  - Centrul Medical Unirea SRL, Brasov
  - Ponderas Academic Hospital, Bucharest
  - Institutul Oncologic Ion Chiricuta, Cluj-Napoca
  - Regina Maria, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Pius Brinzeu, Timișoara
- South Korea (8):
  - Chungbuk National University Hospital, Chungcheongbuk Do
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (9):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Fund. Puigvert, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp.Univ.Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- United Kingdom (4):
  - St Bartholomews Hospital, London
  - Salford Royal Hospital, Salford
  - Southampton University Hospital, Southampton
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency